CLINICAL TRIAL: NCT03731949
Title: Placental Volume Analysis and Monitoring and Vascularity Assessment
Brief Title: Placental Volume Analysis During Pregnanay
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Lecturer, Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: placental growth
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Placenta Diseases
MeSH Terms: conditions — Placenta Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Ultrasonography to assess placental volume

SUMMARY:
Placenta grows with advancing gestational age amonitoring of placental growth is important in pregnancy evaluation

DETAILED DESCRIPTION:
assessment of placental size is very important in evaluating the pregnancy Placenta is one of the most important organs that control pregnancy outcome

ELIGIBILITY:
Inclusion Criteria:

* pregnant ladies between 20 - 40 years old
* ladies pregnant from 14 weeks till term

Exclusion Criteria:

* pregnant ladies in first trimester

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: * pregnant ladies between 20 - 40 years old
  * ladies pregnant from 14 weeks till term
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-05 (Estimated)

PRIMARY OUTCOMES:
the volume of every placenta at the given time of scan | within 2 months
  volume of placenta that will increase with time

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt